CLINICAL TRIAL: NCT06147089
Title: Biomarker Based Intervention Strategies to Combat Adverse Effects of Shift Work
Brief Title: Shift Work Intervention Strategies for Night Shift Workers
Acronym: GRIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: National Institute for Public Health and the Environment (RIVM) (Other Government); Netherlands Organisation for Scientific Research (Other Government)
Responsible Party: Principal Investigator, Dr. Heidi Lammers-van der Holst PhD, Assistant Professor, PhD, Erasmus Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MEC-82649; NL82649.078.22 (Other: Erasmus Medical Center)
Record Dates: First submitted 2023-01-24; First posted 2023-11-27 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Shift-Work Related Sleep Disturbance
Keywords: night shift work; sleep; nutrition; personalised intervention; biomarker; alertness; performance

STUDY DESIGN:
Intervention Model Description: There are three study arms: control group, personalised sleep intervention, and personalised nutritional intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (No Intervention): The control group will receive no behavioral intervention and is instructed to continue with their normal sleep and nutritional habits.
- Sleep intervention (Experimental): The sleep intervention group will receive personalised sleep advice to promote better sleep during night shift periods. This intervention will last 3 months.
  Interventions: Behavioral: Sleep Intervention
- Nutritional Intervention (Experimental): The nutritional intervention group will receive personalised nutrition advice to promote better metabolic health during night shift periods. This intervention will last 3 months.
  Interventions: Behavioral: Nutritional intervention

INTERVENTIONS:
Behavioral: Sleep Intervention — Participants in the sleep intervention receive advice on: sleep hygiene/environment, sleep timing, naps, and exposure to light. These advices will be tailored to the personal situation of the participant, as measured during the run-in period.
  Arms: Sleep intervention
Behavioral: Nutritional intervention — Participants in the nutritional intervention receive personalised advice on the distribution of calories and nutrients over 24 hrs, and on specific food products based on the outcomes of the continuous glucose measurements (CGM) during the run-in period. The guidelines will include room for personal dietary preferences.
  Arms: Nutritional Intervention

SUMMARY:
The goal of this intervention study is to test behavioral interventions in night shift workers. The main question it aims to answer is:

• Can personalized sleep or nutrition intervention strategies help against the negative health effects of night shift work?

Participants will be followed before and after the intervention. Participants will wear smart devices, do a alertness/performance test and complete questionnaires. Blood samples will be collected.

Researchers will compare the intervention groups to the control group (which receives no intervention) to see if the sleep and nutrition interventions affected the health of night shift workers.

DETAILED DESCRIPTION:
Rationale: Night work interferes with the timing of daily activities and disturbs the circadian rhythms of multiple physiological processes in the human body. This is associated with detrimental health effects, such as disturbances in sleep (shorter, less consolidated sleep) and insulin regulation (due to altered eating behaviour). Night shift work is prevalent and difficult to limit in many job types, yet there is currently limited evidence on effective interventions to prevent the health consequence of shift work in a real life context. Therefore more research on tools for the prevention of negative health effects is warranted.

Objective: The current study aims to investigate two types of preventive interventions in night shift workers: a personalised sleep intervention and a personalised nutritional intervention. It will assess the effects of the two interventions on sleep and on (continuous) glucose patterns.

Study design: A non-blinded controlled intervention study, consisting of a run-in period with baseline levels, an intervention of ~ 3 months including measurements at the start of the intervention, a post-intervention measurement and a follow up after 12 months. Study population: The study population consists of employees who work at least 4 night shifts a month on average, with at least 1 year prior experience with shift work. Employees are aged 18-60 years and without a diagnosis of major disease. Each arm of the study will include 25 participants. There are three study arms: control group (no advice), personalised sleep intervention, and personalised nutritional intervention.

Intervention: Participants in the sleep intervention receive advice on: sleep hygiene/environment, sleep timing, naps, and exposure to light. These advices will be tailored to the personal situation of the participant, as measured during the run-in period. Participants in the nutritional intervention receive personalised advice on the distribution of calories and nutrients over 24 hrs, and on specific food products based on the outcomes of the continuous glucose measurements (CGM) during the run-in period. The guidelines will include room for personal dietary preferences. The control group is asked to carry on with their normal sleep and nutritional habits.

Main study parameters/endpoints: The primary outcomes are the quality and quantity of sleep and stability and levels of (continuous) glucose patterns. Secondary outcomes include a set of relevant clinical biomarkers (of metabolic health, epigenetic DNA methylation profiles in blood, and stress markers in hair, and anthropometrics), and alertness during night shifts. For the nutritional intervention, metabolic flexibility and inflammatory resilience will be measured with the mixed-meal challenge test (PhenFlex) test. The outcomes will be compared, pre- and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 60 years.
* Work at least 4 night shifts a month on average.
* Shift workers, working rotating shifts (morning, evening and night shifts) or working predominantly night shifts. Night shift defined as work at least 1 hours between 0:00- and 6:00.
* Work at least 2 night shifts in a row
* Work ≥ 20 work hours per week.
* Having a shift duration of 6 h-12 h.
* History of ≥ 1 year of working rotating shift work or night shifts prior to the study.

Exclusion Criteria:

* Taking medication that the investigator believes would interfere with the objectives of the study. For example, sleep medication, medication that interferes with glucose homeostasis, and/or anti-inflammatory drugs.
* Pregnant or have a wish to become pregnant during the study period.
* Planned surgery during the entire study period Alcohol consumption > 21 units/week
* Severe psychiatric disease and/or any mental or physical disability that will hinder participation in the interventions
* Severe cardiovascular disease, to the discretion of the study doctor
* Having a chronic inflammatory disease, including asthma, rheumatic fever, irritable bowel disease, chronic obstructive pulmonary disease.
* Other bowel diseases, including Chron's disease and Colitis Ulcerosa.
* A disease or condition with higher bleeding risk (/risk of hemorrhage), under which a blood sample may lead to complications.
* Participation in any clinical trial including blood sampling and/or administration of substances up to 90 days before Day 01 of this study
* Recent blood donation (<1 month prior to the start of the study)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Change in Total sleep time (TST) after1 month and 5 months intervention | Baseline, 1 month and 5 months after start intervention
  The TST is calculated as minutes of sleep in the main sleep episode plus the minutes of sleep during any naps between the consecutive shifts, derived from actigraphy data collected in 60 s epochs. The investigators will use a commercial software package to score the sleep.
Change in Fragmentation index (FI) with actigraphy, and calculated using commercial software. Change in Fragmentation Index (FI) after 1 month and 5 months intervention | Baseline, 1 month and 3-5 months after start intervention
  FI will be calculated as the number of times that sleep was terminated after 1 minute, expressed as a percentage of total estimated sleep time, using actigraphy data and commercial software to calculate it.
Change in Wake after sleep onset (WASO) after 1 month and 3-5 months intervention | Baseline, 1 month and 3-5 months after start intervention
  WASO is an objective sleep quality measure and will be calculated as the duration (in minutes) of all awakenings during the main sleep episode measured with actigraphy, and calculated using commercial software.
Change in 24h glucose levels after 1 month and 3-5 months of intervention | Baseline, 1 month and 3-5 months after start intervention
  24h interstitial glucose levels were recorded for 14 days around scheduled transition from day to night shifts, using the Freestyle Libre-Pro.

SECONDARY OUTCOMES:
Change in Subjective Alertness via Karolinska Sleepiness Scale (KSS) after 1 month and 3-5 months of intervention | Baseline, 1 month and 3-5 months after start intervention
  Participants will complete the Karolinska Sleepiness Scale (KSS) as a measure of subjective alertness at the beginning and end of 2 night shifts. The KSS is a Likert scale ranging from 1, extremely alert, to 9, extremely sleepy.beginning and end of 2 consecutive night shifts, to be performed on a mobile phone.
Change in Sustained Attention after 1 month and 3-5 months of intervention | Baseline, 1 month and 3-5 months after start intervention
  The psychomotor vigilance task (PVT) is a test of visual reaction time (RT) in which the participant is asked to maintain the fastest possible RTs to a simple visual stimulus for several minutes. The inter-stimulus interval varies randomly between 2-10 seconds. While there are a number of standard performance metrics that can be obtained from each PVT, we will use the number of lapses of attention (RT > 500msec) as our outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi M Lammers-van der Holst, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van der Rhee M, Oosterman JE, Wopereis S, van der Horst GTJ, Chaves I, Dolle MET, Burdorf A, van Kerkhof LWM, der Holst HML. Personalized sleep and nutritional strategies to combat adverse effects of night shift work: a controlled intervention protocol. BMC Public Health. 2024 Sep 19;24(1):2555. doi: 10.1186/s12889-024-20022-w. PMID 39300419